CLINICAL TRIAL: NCT05917951
Title: Study on Clinical Use of Evusheld (AZD7442) in the Real-world Setting - A Multi-Centre, Single-arm, Observational Study to Determine the Utilisation and Clinical Outcomes of Evusheld in China
Brief Title: Study on Determine the Utilisation and Clinical Outcomes of Evusheld in COVID-19 PrEP in China
Acronym: CLEAR
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8850R00019
Record Dates: First submitted 2022-12-02; First posted 2023-06-26 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evusheld(AZD7442) is a combination of 2 human long-acting antibodies, which was selected for maximal potency and demonstrated synergistic neutralization of SARS-CoV-2 in vitro. PROVENT is a Phase III study in participants at an increased risk for inadequate response to COVID-19 vaccine, an increased risk of exposure to SARS-CoV-2 or both. The study met the primary endpoint of reduction in the incidence of symptomatic Coronavirus disease 2019 (COVID-19) with tixagevimab/cilgavimab (TIXA/CILGA) compared with placebo, risk reduction 76.7% (95% CI, 46.0-90.0), in 5172 patients who did not have a Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) Reverse transcription polymerase chain reaction (RT-PCR) positive COVID-19 infection at baseline. Although the PROVENT trial was invaluable in demonstrating AZD7442's ability to prevent symptomatic infection, it was conducted in highly controlled environments using a rigorous protocol, which does not accurately reflect the patient experience in clinical practice. Furthermore, the sample size of Asian population in phase 3 clinical trials is small (110 subjects in AZD7442 group and 60 subjects in placebo group), and there is very limited clinical trial/real-world data in Chinese population is reported. Therefore, this current study aims to describe the utilisation and clinical outcomes of AZD7442 in Chinese population for pre-exposure prophylaxis.

DETAILED DESCRIPTION:
COVID-19 has a spectrum of clinical manifestations and multisystem organ involvement due to SARS-CoV-2, viral dynamics may correlate to the severity of illness and disease outcomes. Despite the increase in COVID-19 vaccine roll-out, many individuals still remain at high risk of breakthrough infection and many of these individuals are also at higher risk of poor COVID-19 outcomes. In the US about 3% of the adult population is moderately to severely immunocompromised, leading to increased vulnerability to COVID-19.

AZD7442 is a combination of 2 human long acting antibodies, which was selected for maximal potency and demonstrated synergistic neutralization of SARS-CoV-2 in vitro. AZD7442 are 2 monoclonal antibodies that independently neutralize SARS-CoV-2 with high potency in vitro. AZD7442 targets SARS-CoV-2 spike protein to prevent virus entry into host cells.

PROVENT is a Phase III study in participants at an increased risk for inadequate response to COVID-19 vaccine, an increased risk of exposure to SARS-CoV-2 or both. The study met the primary endpoint of reduction in the incidence of symptomatic COVID-19 with TIXA/CILGA compared with placebo, risk reduction 76.7% (95% CI, 46.0-90.0), and longer (median 6-month) follow-up showed a risk reduction of 82.8%, in 5172 patients who did not have a SARS-CoV-2 RT-PCR-positive COVID-19 infection at baseline. Most adverse events were mild or moderate in intensity, with the overall adverse event profile over a median follow-up of 6 months remaining similar to the primary safety analysis. At either the primary or 6-month analyses, there were no cases of severe/critical COVID-19 in those treated with AZD7442. In the placebo arm, there were 5 cases of severe/critical COVID-19 in total.

Although the PROVENT trial was invaluable in demonstrating AZD7442's ability to prevent symptomatic infection, it was conducted in highly controlled environments using a rigorous protocol, which does not accurately reflect the patient experience in clinical practice. Furthermore, the sample size of Asian population in phase 3 clinical trials is small (110 subjects in AZD7442 group and 60 subjects in placebo group), and there is very limited clinical trial/real-world data in Chinese population is reported.

Studies are therefore needed to understand who is being administered AZD7442 in the real world, the frequency of COVID-19 related events, and healthcare resource utilisation (HCRU). Also, important to understand is the potential impact that AZD7442 administration may have on COVID-19 risk behaviours (particularly shielding and other preventive measures), which may in turn influence interpretation of AZD7442 effectiveness results. Such information is imperative to inform clinical decision-making for the care of this relatively vulnerable population.

Therefore, this current study aims to describe the utilisation and clinical outcomes of AZD7442 in Chinese population for pre-exposure prophylaxis. Although this study will not evaluate the effectiveness of AZD7442, the descriptive results may guide further development of studies to assess real world effectiveness of AZD7442. The study is planned to be conducted in approximately 100 sites in China.

ELIGIBILITY:
Inclusion Criteria

Subjects who fulfil all the following inclusion criteria will be eligible to participate in the study:

* Individuals receiving AZD7442 before enrolment date or have been prescribed or have planned to administrate at enrolment date.
* Individuals willing and able to sign informed consent signed.

Exclusion Criteria

Subjects who fulfil any of the following exclusion criteria will not be eligible to participate in the study:

• Individuals currently participating in interventional clinical trials of SARS-CoV-2 prophylactic or treatments.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants included in this this study are all individuals who have received AZD7442 since AZD7442 will be on market in China.
Sampling Method: Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2022-12-24 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
To describe the baseline demographic and clinical characteristics of individuals receiving AZD7442 for pre-exposure prophylaxis | up to 12 months before first administration of AZD7442 for pre-exposure prophylaxis
  * Proportion of individuals by demographic variables of interest (e.g. age, gender, race/ethnicity, smoking status, weight(kg) and height(cm) will be combined to reported body mass index(BMI) in kg/m^2, cities of frequency travel and residence, long-term care or assisted living, household composition, high risk contacts)
  * Proportion of individuals by clinical characteristics of interest (e.g. comorbidities, prior and concurrent medications, including immunosuppressors by type/class)
  * Proportion of individuals by baseline COVID-19 vaccination status or any history of exposure to other prophylactic interventions for prevention of SARS-CoV-2 exposure.
  * Proportion of individuals by baseline history of SARS-CoV-2 infection/COVID-19 diagnosis and disease severity.
  * Proportion of individuals by priority AZD7442 subpopulations of interest

SECONDARY OUTCOMES:
To describe the baseline demographic and clinical characteristics of individuals receiving AZD7442 for pre-exposure prophylaxis by population subgroup of key basic disease. | up to 12 months before first administration of AZD7442 for pre-exposure prophylaxis
  To describe the baseline demographic and clinical characteristics of individuals receiving AZD7442 for pre-exposure prophylaxis by population subgroup of immune compromised disease, including haematological malignancies, solid organ transplant, autoimmune disease, solid tumour, chronic kidney disease (CKD; including dialysis) and others
To describe the incidence of SARS-CoV-2 infection (asymptomatic or symptomatic), medically-attended COVID-19, and COVID-19 related hospitalization and death up to 6 months after first administrationxposure prophylaxis of AZD7442 for pre-e | 6 months after first administration of AZD7442 for pre-exposure prophylaxis
  * Medically attended COVID-19 rate
  * SARS-CoV-2 infection rates (asymptomatic or symptomatic)
  * Proportion of SARS-CoV-2 infection (asymptomatic or symptomatic) in close contacts
  * Proportion of SARS-CoV-2 infection from different cities
  * Type of COVID-19 Variant
  * COVID-19 mortality rates
  * COVID-19 hospitalisation rates
  * COVID-19 intensive care unit (ICU) admission rates
To describe the incidence of all-cause hospitalization and mortality during the 6 months after first administration of AZD7442 for pre-exposure prophylaxis | during the 6 months after first administration of AZD7442 for pre-exposure prophylaxis
  * All cause hospitalisation rate
  * All-cause mortality rate
To describe COVID-19 risk behaviours at the time of AZD7442 injection and during the 6 months after first administration of AZD7442 for pre-exposure prophylaxis | during the 6 months after first administration of AZD7442 for pre-exposure prophylaxis
  • AstraZeneca-developed Risk Behaviour Questionnaire (Appendix A)
To describe COVID-19-related healthcare resource utilisation (HCRU) during the 6 months after first administration of AZD7442 for pre-exposure prophylaxis | during the 6 months after first administration of AZD7442 for pre-exposure prophylaxis
  * Hospitalization, and days hospitalised
  * Supplemental oxygen, and days under supplemental oxygen
  * Re-admission, days in hospital
  * ICU admissions and days in ICU
  * Emergency department (ED) visits
  * Outpatient visits/calls (specialist)
  * COVID-19 related medications or treatment
  * Others
To describe the safety of AZD7442 during the 6 months after first administration of AZD7442 | during the 6 months after first administration of AZD7442 for pre-exposure prophylaxis
  * Serious adverse events (SAEs)
  * Adverse events of special interest (AESIs)
  * Adverse drug reaction (ADR)

OTHER OUTCOMES:
To describe the demographic and clinical characteristics of SARS-CoV-2 infection, medically attended COVID-19, and COVID-19 related hospitalized cases occurring in comparison to non-cases. | 6 months following AZD7442 first administration for pre-exposure prophylaxis
  * Proportion of individuals by demographic variables of interest (e.g. age, gender, race/ethnicity, smoking status, body mass index [BMI, weight in kilograms, height in meters, then weight and height will be combined to reported BMI in kg/m^2], long-term care or assisted living, high risk contacts)
  * Proportion of individuals by clinical characteristics of interest (e.g. comorbidities, prior and concurrent medications, including immunosuppressors by type/class)
  * Proportion of individuals by baseline COVID-19 vaccination status or any history of exposure to other prophylactic interventions for prevention of SARS-CoV-2 exposure
  * Proportion of individuals by baseline history of SARS-CoV-2 infection/COVID-19 diagnosis and disease severity
  * Proportion of individuals by priority AZD7442 subpopulations of interest
To describe the incidence of long COVID syndrome following AZD7442 first administration for pre-exposure prophylaxis | 12 weeks from first onset of COVID-19 symptoms
  * Proportion of subjects with long-COVID syndrome at >12 weeks from first onset of COVID-19 symptoms
  * Duration of long COVID syndrome: medium (days, interquartile range (IQR), minimum, maximum; and mean standard deviation)
To describe the baseline and repeat administration(s) of AZD7442 | when receive AZD7442
  Number, frequency of subjects administered AZD7442 by:
  * Route of administration (e.g. IM or IV)
  * Dose number, location (e.g. thigh or gluteus), amount and timing/interval between doses o Type of medical condition
To describe the usage purpose of AZD7442 | when receive AZD7442
  Number, proportion of subjects administered AZD7442 by:
  * Pre-exposure Prophylaxis
  * Post-exposure Prophylaxis
  * Treatment of mild/Asymptomatic disease
  * Treatment of normal disease
  * Treatment of severe disease
To describe SARS-CoV-2 RNA viral load levelsafter symptomatic SARS-CoV-2 infection within 29 days after first administration of AZD7442 for treatment | within 29 days after first administration of AZD7442 for treatment
  • SARS-CoV-2 RNA viral load levels and changes in nasal swabs during hospitalization up to 29 days
To describe the neutralising responses against SARS-CoV-2 subvariants of AZD7442 in serum (if applicable) | 6 months following AZD7442 first administration for pre-exposure prophylaxis
  • Post treatment GMTs and GMFRs from baseline value through 6 month after single IM dose in SARS-COV-2 neutralizing antibodies (pseudo neutralization assay)
To describe severe COVID-19 related hospitalization and ICU after symptomatic SARS-CoV-2 infection within 29 days after first administration of AZD7442 for treatment | within 29 days after first administration of AZD7442 for treatment
  * Severe COVID-19 hospitalisation rates and days
  * COVID-19 intensive care unit (ICU) admission rates

CONTACTS AND LOCATIONS:
Overall Officials: Jieming Qu, Doctor, Principal Investigator — 18917762988
Locations (1):
- (2) Ruijin-Hainan Hospital Shanghai Jiaotong University School of Medicine (Hainan Boao Research Hospital), Qionghai, Hainan, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for Individual participant data(IPD), but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the European Federation of Pharmaceutical Industries Associations (EFPIA) Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] You J, Wu H, Tian J, Wen J, Shi W, Wang Z, Du Y, Xu H, Wei H, Li X, Kang W, Zhou M, Gu Z, Qu J. Real-world clinical outcomes of tixagevimab/cilgavimab in the Omicron outbreak in China: baseline characteristics and interim analysis of the CLEAR study. Virol J. 2024 Oct 24;21(1):262. doi: 10.1186/s12985-024-02509-5. PMID 39448986
- See also: redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8850R00019&attachmentIdentifier=fd3d7d88-a7af-467b-9d9a-99e692f5c5e9&fileName=D8850R00019_study_report_synopsis.pdf&versionIdentifier=